CLINICAL TRIAL: NCT07110376
Title: Deep Brain Stimulation Neural Recordings of Varied Stimulation During Sleep in Parkinson's Disease - The DREAMS-PD Study
Brief Title: Deep Brain Stimulation Neural Recordings of Varied Stimulation During Sleep in Parkinson's Disease
Acronym: DREAMS-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Parkinson's Disease Association, Inc (Other); Beacon Biosignals (Industry)
Responsible Party: Principal Investigator, James Liao, Staff Physician, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-323 DREAMS-PD
Record Dates: First submitted 2025-07-28; First posted 2025-08-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluate the Impact of Deep Brain Stimulation Settings on Sleep (Experimental): Participants with Parkinson's disease implanted with a Medtronic Percept™ deep brain stimulation (DBS) system will undergo a 6-week in-home monitoring protocol. Each participant will be exposed to three different nighttime-only DBS stimulation settings in a randomized 2-week crossover design: (1) no stimulation (0% amplitude), (2) reduced stimulation (50% amplitude), and (3) optimal clinical stimulation. Sleep metrics will be collected nightly using the Dreem Headband wearable electroencephalogram (EEG) device. One night of polysomnography will also be conducted to validate the wearable. Subcortical local field potentials (LFPs) from the subthalamic nucleus will be recorded to assess band power and coherence during different stimulation settings and sleep stages. The study aims to evaluate the effect of DBS settings on sleep efficiency, spectral features of neural activity, and their correlation.
  Interventions: Other: Nighttime Deep Brain Stimulation with Varying Amplitude Settings

INTERVENTIONS:
Other: Nighttime Deep Brain Stimulation with Varying Amplitude Settings — Participants will undergo three different nighttime-only Deep Brain Stimulation (DBS) settings in a randomized crossover design: 0% amplitude (stimulation off), 50% amplitude of their optimal clinical DBS settings, and full clinical DBS settings (100%). Each setting is applied for two weeks during sleep, over a total six-week home monitoring period. The intervention is designed to assess how varying levels of subthalamic nucleus DBS influence sleep quality and neural oscillatory activity. Only nighttime DBS settings are modified; daytime settings remain unchanged.
  Other Names: Nocturnal DBS Amplitude Modulation; DBS Sleep Modulation Protocol; 0%, 50%, 100% DBS Night Settings

SUMMARY:
This study employs an exploratory, prospective, single center, naturalistic clinical trial design with a randomized crossover intervention.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) stands as an established and robust treatment for various motor symptoms in patients with Parkinson's disease (PWP). While it has shown promise in ameliorating non-motor symptoms, the mechanisms underlying these improvements remain poorly understood. A significant forthcoming shift in the DBS landscape is the transition towards closed-loop or "adaptive DBS" (aDBS). This approach relies on expanding knowledge of basal ganglia electrophysiology and its correlation with motor symptoms. Augmented beta frequency oscillations (13-35 Hz) in local field potentials (LFP) from the basal ganglia is correlated with severity of the motor systems bradykinesia/rigidity and serve as an electrophysiological biomarker for clinical state. Essentially, aDBS aims to modulate stimulation in response to neural state, offering more precise symptom control.

Sleep disturbances are a prevalent symptom in PWP, affecting a vast majority of patients, and serve as a significant non-motor contributor to quality of life. While DBS has demonstrated benefits in enhancing sleep efficiency and architecture, the mechanisms by which this might occur, as well as the optimal stimulation parameters for treating sleep dysfunctions are unknown. Sleep is associated with a dramatic change in subcortical neural activity compared to the wake state, with decreased beta activity, which could serve as a neurophysiological biomarker for the sleep state. Since beta frequencies are a common target for adaptive DBS studies in PD, addressing sleep-induced reductions in beta activity will be crucial for future algorithm development. Incorrectly interpreting sleep as the "medication-on" state may result in an adaptive algorithm providing the patient with non-optimal stimulation amplitudes that may adversely affect sleep.

There is an urgent need to identify the dose-response curve regarding how stimulation affects sleep quality and neurophysiology. Our primary objective is to address this knowledge gap by obtaining a comprehensive understanding of the subcortical neural signatures of sleep, and their correlation with sleep outcomes under different stimulation currents. This will ultimately enable us to establish the control policy for adaptive control of stimulation amplitude (current). Our central hypothesis is that different stimulation currents will elicit distinct effects on sleep subcortical neural signatures and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age
* Diagnosed with idiopathic Parkinson Disease
* Have bilateral implantation of Medtronic's PerceptTM PC (Medtronic Neurological Division, Minneapolis, MN, USA) Deep Brain Stimulation (DBS) system targeting the subthalamic nucleus (STN) and have had their stimulation settings optimized for a minimum of three months
* Report a response score of one or greater on question 1.7 of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part I;
* Demonstrate ability to ambulate independently;
* Be capable of providing informed consent;
* If taking sleep-supporting medications, dosing must be stable for at least 30 days

Exclusion Criteria:

* Presence of neurological diseases other than Parkinson Disease, such as stroke or multiple sclerosis
* Active sleep disorders, including narcolepsy, moderate to severe (Apnea-Hypopnea Index>=15) untreated sleep apnea, uncontrolled restless legs syndrome
* Cognitive impairment meeting the criteria for dementia as per the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV), based on formal neuropsychological evaluation
* Ongoing alcohol or substance abuse; Working night shifts or irregular work hours

The main concern for vulnerable subjects will be for the possibility of reduced decision-making capacity. For this we intend to exclude individuals who have a diagnosis of dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To demonstrate differences in sleep efficiency (SE) among different stimulation settings. | At the end of each 2-week stimulation period (over 6 weeks total)
  Sleep efficiency will be calculated as: (total sleep time ÷ total time in bed) × 100, using nightly data collected via the Dreem Headband. The mean SE for each 2-week stimulation setting (0%, 50%, 100% amplitude) will be compared within subjects using crossover analysis.

SECONDARY OUTCOMES:
Average Nightly Beta Band Power | At the end of each 2-week stimulation period (over 6 weeks total)
  Average beta band power will be derived from subthalamic nucleus local field potentials recorded via the Medtronic Percept™ system.
Correlation Between Sleep Efficiency and Beta Band Power | Over each night during the 6-week study period
  The correlation between sleep efficiency (measured by Dreem Headband) and beta band power (recorded from DBS electrodes) will be evaluated. Analyses will include full-night averages and specific sleep stages (N1/N2, N3).
Correlation of Wake After Sleep Onset (WASO) with Beta Band Power | Across 6-week study period and at the end of each 2-week stimulation phase
  Wake after sleep onset (WASO) will be analyzed in relation to Deep Brain Stimulation (DBS) band power. Relationships will be examined across each stimulation condition and averaged over the study.
Coherence Across Deep Brain Stimulation Amplitude Settings | At the end of each 2-week stimulation period (over 6 weeks total)
  Coherence between left and right subthalamic nucleus (STN) will be calculated. Comparisons will be made across the three stimulation settings
Correlation of sleep fragmentation index with Beta Band Power | Across 6-week study period and at the end of each 2-week stimulation phase
  Sleep fragmentation index will be analyzed in relation to Deep Brain Stimulation (DBS) band power. Relationships will be examined across each stimulation condition and averaged over the study.
Correlation of Pittsburgh Sleep Quality Index (PSQI) with Beta Band Power | Across 6-week study period and at the end of each 2-week stimulation phase
  Pittsburgh Sleep Quality Index (PSQI) will be analyzed in relation to Deep Brain Stimulation (DBS) band power. Relationships will be examined across each stimulation condition and averaged over the study.
Correlation of and Epworth Sleepiness Scale (ESS) with Beta Band Power | Across 6-week study period and at the end of each 2-week stimulation phase
  Epworth Sleepiness Scale (ESS) will be analyzed in relation to Deep Brain Stimulation (DBS) band power. Relationships will be examined across each stimulation condition and averaged over the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States